CLINICAL TRIAL: NCT06285513
Title: Metabolic Remodeling Assessment During Severe Cardiovascular Dysfunction in Shock
Brief Title: Cardiovascular Metabolic Remodeling in Shock
Acronym: METASHOCK
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/387/OB; 2023-A00503-42 (Registry Identifier: Frecnh Ministry)
Record Dates: First submitted 2024-01-02; First posted 2024-02-29 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2023-12

CONDITIONS: Shock
Keywords: Metabolic remodelling; Shock states; Cardiovascular dysfunction; Metabolomics
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Diagnostic Test: Cardiac ultrasound — Cardiac ultrasound : determination of impairment of cardiac function by echocardiographic analysis (at V1, V3 and V4), Glycocheck : automatic analysis of sublingual microcirculation, Indirect calorimetry : determining the increase in energy expenditure in patients with septic shock
  Other Names: GlycoCheck; Indirect calorimetry (in case of artificial ventilation)

SUMMARY:
The aim of the study is to increase our knowledge of energy dysfunction in the cardiovascular dysfunction observed during shock states by analysing the omics molecules involved.

DETAILED DESCRIPTION:
To do this, the investigators chose to carry out an in-depth study of the different metabolic pathways, using metabolomic analysis of plasma, targeting the cardiovascular metabolism of patients admitted to intensive care for septic and non-septic shocks.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 18 and 75.
* Patient admitted to intensive care for shock treated with a vasoactive or inotropic amine (adrenaline, dobutamine or noradrenaline).Patient undergoing invasive mechanical ventilation for less than 24 hours (or admitted to intensive care for less than 24 hours if the patient arrived intubated) and for a foreseeable duration of ventilation of at least 48 hours.
* Patient, or relative if the patient is not competent, who has read and understood the information letter and does not object to participation in the research, or emergency procedure in the absence of a relative.
* Urine or blood pregnancy test if a sample is taken as part of routine negative care (if woman of childbearing age).

Exclusion Criteria:

* Moribund patient (death expected within < 24 hours) and/or decision to limit or stop treatment on admission to intensive care.
* Pregnant, parturient or breast-feeding woman.
* Patient not suitable for enteral calorie intake. Patient with a history of: advanced chronic renal failure ; advanced chronic liver failure.
* Incapacitated patient of full age (under guardianship, curatorship) or deprived of liberty by court order.
* Patient already taking part in an interventional study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalised in intensive care for shock, treated with a vasoactive or ionotropic amine, undergoing invasive mechanical ventilation for less than 24 hours
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the prognostic capacity of the initial metabolomic profile of patients in shock | Day 3
  Correlation between plasma concentrations of metabolites at inclusion and delta of SOFA score (SOFA Day 1 - SOFA Day 3) with adjustment for SOFA at Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire JOLLY, MD, Principal Investigator — University Hospital of Rouen, France
Locations (1):
- University Hospital of Rouen, Rouen, France

IPD SHARING:
Plan to Share IPD: No